CLINICAL TRIAL: NCT06961812
Title: Validation of the Self-Assessment for Falls in the Elderly (SAFE) Questionnaire to Assess the Risk of Falls in People Aged 60 or Over.
Acronym: SAFE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: REHCMPL25_0035
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Fall Prevention; Falls (Accidents) in Old Age
Keywords: Falls; Functional Assessment; Predictive Value of Tests; Aging; Fallers Aged 60 Years and Older
MeSH Terms: interventions — Physical Examination

STUDY DESIGN:
Intervention Model Description: single-centre, cross-sectional diagnostic
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fall Risk Assessment (Experimental): Patients or carers over 60 consulting the geriatrics department at Montpellier University Hospital
  Interventions: Diagnostic Test: Questionnaire and Physical Exam; Diagnostic Test: Safe Self-Administered Questionnaire

INTERVENTIONS:
Diagnostic Test: Questionnaire and Physical Exam — Next, the risk of falling will be assessed by a healthcare professional using a hetero-questionnaire and physical tests, as proposed in the algorithm for global recommendations (routine care).
  These tests include a detailed characterisation of the history of falls, the Timed Up and Go, the Five Times Sit to Stand, the 4 m walking speed and the Short Physical Performance Battery.
Diagnostic Test: Safe Self-Administered Questionnaire — All people who agree to take part in the study will first complete the SAFE self-questionnaire (intervention).
  the Self Assessment for Falls in the Elderly (SAFE), an auto-questionnaire that converts the binary items and performance tests of the 2022 World Guidelines for Falls Prevention and Management into visual analogue scales (100 mm each).

SUMMARY:
This single-centre, cross-sectional diagnostic study will determine whether the new self-completed Self-Assessment for Falls in the Elderly (SAFE) questionnaire can classify fall-risk level (low, moderate, high) in adults ≥ 60 years as accurately as the current clinician-administered international algorithm that mixes yes/no questions with physical tests; to do so, about 300 participants will (1) sign consent, (2) answer the 5-minute SAFE, and (3) undergo guideline assessment and tests by a clinician in the same visit, after which researchers will compare SAFE and clinician results for sensitivity, specificity, and predictive values, examine agreement and correlations, and give immediate risk-based prevention advice:

* Eligibility: men or women ≥ 60 y, stable walking/balance ≥ 1 month, able to read French and perform brief tests; legal guardianship or refusal excludes.
* Participant tasks: complete SAFE; perform Timed Up-and-Go, 4 m gait speed, Five-Times-Sit-to-Stand and Short Physical Performance Battery (SPPB) under supervision
* Benefits/Risks: instant personalised fall-risk feedback; SAFE is risk-free and physical tests carry only minimal supervised exertion.

Falls are a leading cause of injury and death in older adults, and current assessments require trained staff; if SAFE proves equivalent, it could enable large-scale, low-cost self-screening and support future digital monitoring tools for fall prevention.

DETAILED DESCRIPTION:
This single centre diagnostic accuracy study validates the Self Assessment for Falls in the Elderly (SAFE), an auto-questionnaire that converts the binary items and performance tests of the 2022 World Guidelines for Falls Prevention and Management into visual analogue scales (100 mm each). SAFE is completed without assistance in ≈ 5 min and yields a continuous score that can be stratified into low, moderate, or high fall risk categories. The reference standard is the full guideline algorithm-Three Key Questions, detailed fall history characterisation, Timed Up and Go, Five Times Sit to Stand, 4 m gait speed, and Short Physical Performance Battery-administered by a trained clinician after the participant has returned the SAFE form to prevent incorporation bias.

The study adopts a cross sectional design and will recruit 300 community dwelling adults aged ≥ 60 years attending the Geriatrics Department of Montpellier University Hospital over 6 months. Sample size (300) was calculated for expected sensitivity and specificity of 0.85, 30 % prevalence of moderate to high fall risk, 5 % absolute precision, two sided α = 0.05, and 90 % power. After informed consent and eligibility verification, participants complete a single study visit in the following order: (1) SAFE self completion, (2) guideline interview plus physical tests. No investigational product, device, imaging, or biospecimen collection is involved.

Statistical plan. For every SAFE VAS (visual analogue scale) item, optimal cut points will be derived from non parametric ROC analysis versus its binary analogue. The primary analysis compares the three level SAFE classification with the reference standard using contingency tables and reports sensitivity, specificity, positive and negative predictive values, likelihood ratios, diagnostic odds ratio, and area under the summary ROC curve with 95 % confidence intervals. Secondary analyses will explore Pearson or point biserial correlations between individual SAFE scores and continuous physical test results, apply multivariable ordinal logistic regression to evaluate whether age, sex, or comorbidity modify SAFE performance, and perform decision curve analysis to estimate net clinical benefit across plausible threshold probabilities. Missing data will be handled by complete case analysis.

Data quality and monitoring. Source data will be captured in an electronic case report form with automated range and consistency checks. The CHU Montpellier sponsor will conduct risk based on site and/or remote monitoring and centralised statistical data surveillance. All study documentation will be archived for 15 years in line with French regulations.

Ethics, safety, and dissemination. The protocol has been submitted to a French Comité de Protection des Personnes and the Agence Nationale de Sécurité du Médicament (category 3). Physical testing is performed by certified staff in a dedicated fall prevention clinic with immediate assistance available; adverse events are therefore not expected but will be recorded and reported according to Good Clinical Practice. Results-positive, negative, or inconclusive-will be published in peer reviewed journals and communicated to participants on request. Should SAFE demonstrate acceptable diagnostic accuracy, its simplicity will enable large scale, low cost self screening, integration into mobile health applications, and targeted allocation of fall prevention resources for older adults.

ELIGIBILITY:
Inclusion Criteria:

* People aged 60 or over, judged by the investigator to be in stable clinical condition as regards walking and balance for at least one month,
* Able to perform the necessary physical assessments

Exclusion Criteria:

* Unable, according to the investigator, to answer a self-questionnaire,
* Patient's refusal to take part in the study
* Absence of a caregiver if the participant is unable to answer the questionnaire alone
* Unable to understand the information note
* Opposition of the proxy or legal guardian if the participant is under legal protection (guardianship, curatorship, safeguard of justice)
* Subject deprived of liberty (art. L. 1121-6) (by judicial or administrative decision, or forced hospitalization)
* Not affiliated to a French social security scheme or beneficiary of such a scheme (L1121-8-1)
* Participation in other research involving a period of exclusion still in progress (Article L1121-12)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-05-02 (Estimated); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Performance of the SAFE Self-Assessment Questionnaire compared with the global recommendations algorithm (Hetero-administered questionnaire and physical tests). sensitivity | At inclusion
  Based on predefined VAS thresholds in the self-questionnaire, we apply the global recommendations algorithm to classify patients into low, moderate, and high risk of falling:
  High Risk: At least one of the following:
  Two or more falls in the last year. One fall with injury in the last year. One fall with inability to get up in the last year. Unexplained fall in the last year. Frailty: At least three of the five Fried factors (fatigue, >5 seconds for 4 meters, >15 seconds for 5 chair lifts, >4.5 kg weight loss in one year, sedentary lifestyle).
  Moderate Risk: Non-severe fall, fear of falling, or instability while walking/standing, associated with: TUG ≥ 15 seconds, or ≥ 5 seconds to walk 4 meters.
  Low Risk: One non-severe fall, fear of falling, or instability, but no frailty and normal TUG (Timed Up and Go) and walking speed.
  We compare the statistical performance of SAFE with the reference standard using contingency tables, reporting sensitivity
Performance of the SAFE Self-Assessment Questionnaire compared with the global recommendations algorithm (Hetero-administered questionnaire and physical tests). specificity | At inclusion
  Based on predefined VAS thresholds in the self-questionnaire, we apply the global recommendations algorithm to classify patients into low, moderate, and high risk of falling:
  High Risk: At least one of the following:
  Two or more falls in the last year. One fall with injury in the last year. One fall with inability to get up in the last year. Unexplained fall in the last year. Frailty: At least three of the five Fried factors (fatigue, >5 seconds for 4 meters, >15 seconds for 5 chair lifts, >4.5 kg weight loss in one year, sedentary lifestyle).
  Moderate Risk: Non-severe fall, fear of falling, or instability while walking/standing, associated with: TUG ≥ 15 seconds, or ≥ 5 seconds to walk 4 meters.
  Low Risk: One non-severe fall, fear of falling, or instability, but no frailty and normal TUG and walking speed.
  We compare the statistical performance of SAFE with the reference standard using contingency tables, reporting specificity
Performance of the SAFE Self-Assessment Questionnaire compared with the global recommendations algorithm (Hetero-administered questionnaire and physical tests). positive predictive values | At inclusion
  Based on predefined VAS thresholds in the self-questionnaire, we apply the global recommendations algorithm to classify patients into low, moderate, and high risk of falling:
  High Risk: At least one of the following:
  Two or more falls in the last year. One fall with injury in the last year. One fall with inability to get up in the last year. Unexplained fall in the last year. Frailty: At least three of the five Fried factors (fatigue, >5 seconds for 4 meters, >15 seconds for 5 chair lifts, >4.5 kg weight loss in one year, sedentary lifestyle).
  Moderate Risk: Non-severe fall, fear of falling, or instability while walking/standing, associated with: TUG ≥ 15 seconds, or ≥ 5 seconds to walk 4 meters.
  Low Risk: One non-severe fall, fear of falling, or instability, but no frailty and normal TUG and walking speed.
  We compare the statistical performance of SAFE with the reference standard using contingency tables, reporting positive predictive values,
Performance of the SAFE Self-Assessment Questionnaire compared with the global recommendations algorithm (Hetero-administered questionnaire and physical tests). negative predictive values | At inclusion
  Based on predefined VAS thresholds in the self-questionnaire, we apply the global recommendations algorithm to classify patients into low, moderate, and high risk of falling:
  High Risk: At least one of the following:
  Two or more falls in the last year. One fall with injury in the last year. One fall with inability to get up in the last year. Unexplained fall in the last year. Frailty: At least three of the five Fried factors (fatigue, >5 seconds for 4 meters, >15 seconds for 5 chair lifts, >4.5 kg weight loss in one year, sedentary lifestyle).
  Moderate Risk: Non-severe fall, fear of falling, or instability while walking/standing, associated with: TUG ≥ 15 seconds, or ≥ 5 seconds to walk 4 meters.
  Low Risk: One non-severe fall, fear of falling, or instability, but no frailty and normal TUG and walking speed.
  We compare the statistical performance of SAFE with the reference standard using contingency tables, reporting negative predictive values
Performance of the SAFE Self-Assessment Questionnaire compared with the global recommendations algorithm (Hetero-administered questionnaire and physical tests). likelihood ratios | At inclusion
  Based on predefined VAS thresholds in the self-questionnaire, we apply the global recommendations algorithm to classify patients into low, moderate, and high risk of falling:
  High Risk: At least one of the following:
  Two or more falls in the last year. One fall with injury in the last year. One fall with inability to get up in the last year. Unexplained fall in the last year. Frailty: At least three of the five Fried factors (fatigue, >5 seconds for 4 meters, >15 seconds for 5 chair lifts, >4.5 kg weight loss in one year, sedentary lifestyle).
  Moderate Risk: Non-severe fall, fear of falling, or instability while walking/standing, associated with: TUG ≥ 15 seconds, or ≥ 5 seconds to walk 4 meters.
  Low Risk: One non-severe fall, fear of falling, or instability, but no frailty and normal TUG and walking speed.
  We compare the statistical performance of SAFE with the reference standard using contingency tables, reporting likelihood ratios
Performance of the SAFE Self-Assessment Questionnaire compared with the global recommendations algorithm (Hetero-administered questionnaire and physical tests). diagnostic odds ratio | At inclusion
  Based on predefined VAS thresholds in the self-questionnaire, we apply the global recommendations algorithm to classify patients into low, moderate, and high risk of falling:
  High Risk: At least one of the following:
  Two or more falls in the last year. One fall with injury in the last year. One fall with inability to get up in the last year. Unexplained fall in the last year. Frailty: At least three of the five Fried factors (fatigue, >5 seconds for 4 meters, >15 seconds for 5 chair lifts, >4.5 kg weight loss in one year, sedentary lifestyle).
  Moderate Risk: Non-severe fall, fear of falling, or instability while walking/standing, associated with: TUG ≥ 15 seconds, or ≥ 5 seconds to walk 4 meters.
  Low Risk: One non-severe fall, fear of falling, or instability, but no frailty and normal TUG and walking speed.
  We compare the statistical performance of SAFE with the reference standard using contingency tables, reporting diagnostic odds ratio

SECONDARY OUTCOMES:
VAS thresholds for the self-questionnaire | At inclusion
  In this section, for each binary question on the hetero-questionnaire or involving a physical test, we aim to determine a VAS threshold from the self-questionnaire for the corresponding question. The hetero-questionnaire measure is used as a reference measure: fear of falling, unsteadiness when standing up, unsteadiness when walking, getting up easily from a chair without using hands, walking speed, fatigue, reduction in physical activity.
Concordance analyses | At inclusion
  We wish to evaluate the concordance between the SAFE self-questionnaire responses and the global recommendations algorithm hetero-assessment via the Gwet coefficient for qualitative variables and the intra-class correlation coefficient (ICC) for quantitative variables.
Point-biserial correlations | At inclusion
  We wish to evaluate the correlation between the VAS of the self-questionnaire and the dichotomous variables of the hetero-questionnaire (point-biserial correlations).
Pearson correlation analysis | At inclusion
  We wish to evaluate the correlation between the VAS of the self-questionnaire and the physical tests of the hetero-questionnaire (Pearson correlations).

CONTACTS AND LOCATIONS:
Overall Officials: Jean Baptiste ROBIAUD, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montero-Odasso M, van der Velde N, Martin FC, Petrovic M, Tan MP, Ryg J, Aguilar-Navarro S, Alexander NB, Becker C, Blain H, Bourke R, Cameron ID, Camicioli R, Clemson L, Close J, Delbaere K, Duan L, Duque G, Dyer SM, Freiberger E, Ganz DA, Gomez F, Hausdorff JM, Hogan DB, Hunter SMW, Jauregui JR, Kamkar N, Kenny RA, Lamb SE, Latham NK, Lipsitz LA, Liu-Ambrose T, Logan P, Lord SR, Mallet L, Marsh D, Milisen K, Moctezuma-Gallegos R, Morris ME, Nieuwboer A, Perracini MR, Pieruccini-Faria F, Pighills A, Said C, Sejdic E, Sherrington C, Skelton DA, Dsouza S, Speechley M, Stark S, Todd C, Troen BR, van der Cammen T, Verghese J, Vlaeyen E, Watt JA, Masud T; Task Force on Global Guidelines for Falls in Older Adults. World guidelines for falls prevention and management for older adults: a global initiative. Age Ageing. 2022 Sep 2;51(9):afac205. doi: 10.1093/ageing/afac205. PMID 36178003
- [Background] Montero-Odasso MM, Kamkar N, Pieruccini-Faria F, Osman A, Sarquis-Adamson Y, Close J, Hogan DB, Hunter SW, Kenny RA, Lipsitz LA, Lord SR, Madden KM, Petrovic M, Ryg J, Speechley M, Sultana M, Tan MP, van der Velde N, Verghese J, Masud T; Task Force on Global Guidelines for Falls in Older Adults. Evaluation of Clinical Practice Guidelines on Fall Prevention and Management for Older Adults: A Systematic Review. JAMA Netw Open. 2021 Dec 1;4(12):e2138911. doi: 10.1001/jamanetworkopen.2021.38911. PMID 34910151
- [Background] Ganz DA, Bao Y, Shekelle PG, Rubenstein LZ. Will my patient fall? JAMA. 2007 Jan 3;297(1):77-86. doi: 10.1001/jama.297.1.77. PMID 17200478
- [Background] Park SH. Tools for assessing fall risk in the elderly: a systematic review and meta-analysis. Aging Clin Exp Res. 2018 Jan;30(1):1-16. doi: 10.1007/s40520-017-0749-0. Epub 2017 Apr 3. PMID 28374345
- [Background] Burns ER, Lee R, Hodge SE, Pineau VJ, Welch B, Zhu M. Validation and comparison of fall screening tools for predicting future falls among older adults. Arch Gerontol Geriatr. 2022 Jul-Aug;101:104713. doi: 10.1016/j.archger.2022.104713. Epub 2022 Apr 30. PMID 35526339
- [Background] Blain H, Annweiler C, Berrut G, Becker C, Bernard PL, Bousquet J, Dargent-Molina P, Friocourt P, Martin FC, Masud T, Petrovic M, Puisieux F, Robiaud JB, Ryg J, Van der Velde N, Montero-Odasso M, Rolland Y. [Synthesis in French of the 2022 global recommendations for the management and prevention of falls in the elderly]. Geriatr Psychol Neuropsychiatr Vieil. 2023 Jun 1;21(2):149-160. doi: 10.1684/pnv.2023.1108. French. PMID 37519073
- [Background] Blain H, Annweiler C, Berrut G, Bernard PL, Bousquet J, Dargent-Molina P, Friocourt P, Puisieux F, Robiaud JB, Rolland Y. [Anti-fall plan for the elderly in France 2022-2024: objectives and methodology]. Geriatr Psychol Neuropsychiatr Vieil. 2023 Sep 1;21(3):286-294. doi: 10.1684/pnv.2023.1122. French. PMID 38093564
- [Background] Gillespie LD, Robertson MC, Gillespie WJ, Sherrington C, Gates S, Clemson LM, Lamb SE. Interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD007146. doi: 10.1002/14651858.CD007146.pub3. PMID 22972103
- [Background] Kendrick D, Kumar A, Carpenter H, Zijlstra GA, Skelton DA, Cook JR, Stevens Z, Belcher CM, Haworth D, Gawler SJ, Gage H, Masud T, Bowling A, Pearl M, Morris RW, Iliffe S, Delbaere K. Exercise for reducing fear of falling in older people living in the community. Cochrane Database Syst Rev. 2014 Nov 28;2014(11):CD009848. doi: 10.1002/14651858.CD009848.pub2. PMID 25432016